CLINICAL TRIAL: NCT04644913
Title: Long-term Evaluation of the Quality of Life and the Functional Repercussions of Former Patients Treated With Orthopedic Surgery, With or Without Radiotherapy
Brief Title: Long-term Evaluation of the Quality of Life of Former Patients Treated With Orthopedic Surgery, With or Without Radiotherapy
Acronym: STARTos
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Osteosarcoma in Children
Keywords: Quality of life; Long term follow up; Orthopedic surgery; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Quality of life questionnaire — Sending of 2 questionnaires (SF 36 and TESS)

SUMMARY:
Surgery and radiation therapy play a major role in the treatment of bone and soft tissue tumors. Osteosarcomas, rhabdomyosarcomas, and Ewing tumors are the most common histologic types. Surgery may require multiple techniques and radiation therapy may be conformational, or more recently IMRT (Intensity Modulated Radiation Therapy). If surgery is possible, lower limb surgery is generally the recommended treatment, even if a poor functional result can be expected.

The literature is very poor regarding the impact of radiotherapy on quality of life and functional results, mainly with the use of prosthetic materials.

Tools such as the Toronto Extremity Salvage Score (TESS) are now available for self-assessment of functional outcomes. The presence of large cohorts such as FCCSS, COHOPER and SALTO facilitates these studies.

The SF-36 is a short 36-question health questionnaire that consists of a generic, consistent, and easy-to-administer set of measures. These measures are based on self-report by patients and are now widely used by organizations managing the care of adult patients.

The TESS Functional Questionnaire is a patient-completed self-questionnaire widely used for motor stimulation in patients with musculoskeletal tumors. This score is based on the definitions of handicap, impairment and handicap as documented by the World Health Organization (WHO). It includes 30 questions assessing overall function and daily activities. The final score varies from 0% to 100%, 100% being the best possible score. So far, several studies have reported the validation of TESS in Portuguese, Danish, Korean, Japanese and since this year in French. Indeed, the TESS questionnaire was validated in French by the study "Transcultural validation of TESS and MSTS questionnaires" promoted by the Nantes University Hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients from the French FCCSS or COHOPER or SALTO cohorts Adult patient (> 18 years old) when filling out the study questionnaires Patient treated for a bone tumor before the age of 18 Patient with a minimum follow-up of 5 years without cancer treatment (treated before 2014) Patient living in France and speaking French

Exclusion Criteria:

Patient with a 2nd cancer Patient who has already been approached by the Hospital de NANTES as part of the cross-cultural validation of the TESS questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The PAIR Pediatrics 2017 START project is interested in adults treated for a tumor or malignant hemopathy before the age of 18, in France, since 1980, and with a minimum follow-up of 5 years without cancer treatment.
  The START-os study sample will select patients with at least 5 years of follow-up after childhood sarcoma treated by surgery with or without radiotherapy from the French Childhood Cancer Registry (FCCSS cohorts (patients treated before 2000), COHOPER (patients treated since 2000) and SALTO (patients diagnosed between 1987 and 1992)).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
The concordance of scores from the quality of life questionnaires: SF 36 and TESS | 12 months
  Scoring of questionnaires SF36 and TESS

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane SUPIOT, PHD-MD, Study Director — ICO
Locations (1):
- Institut de Canérologie de l'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No